CLINICAL TRIAL: NCT06703476
Title: A Clinically Integrated Randomized Clinical Trial (RCT) of Modifications to Radical Cystectomy and Postoperative Care
Brief Title: A Study of Surgical Techniques During Cystectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 24-361
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer
Keywords: Cystectomy; Ureteral stents; Alvimopan; 24-361
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — alvimopan

STUDY DESIGN:
Intervention Model Description: This study will use a cluster randomized trial design with crossover wherein surgeons will be cluster randomized for periods of 3 months to use or not use stents and to administer or not administer alvimopan. In addition, a factorial design will be used wherein the 2 study interventions (use of stents and use of alvimopan) will be investigated in the same group of patients.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stent vs No Stent (Experimental): For patients treated by a surgeon randomized to use ureteral stents, the operating surgeon may choose to use a single or double J ureteral stent (6- to 8.5-fr in size) or an alternative ureteral stent of the surgeon's choice to be placed across the ureteroenteric anastomosis intraoperatively. Because there is no standard ureteral stent size or type, the surgeon will select a stent type and size according to their experience and will document the stent size and type used. This is already routinely recorded as part of the standard of care at MSK.
  Interventions: Procedure: Stent placement
- Alvimopan vs No Alvimopan (Experimental): For patients randomized to receive alvimopan, the patient will receive alvimopan as a fixed 12-mg dose, with the first dose administered 0.5 to 5 h before the start of surgery; administration will be continued with twice daily oral doses postoperatively until hospital discharge or a maximum of 7 days (15 in-hospital doses), as indicated on the medication's FDA label. This is the current standard of care for most cases at MSK.
  Interventions: Drug: Alvimopan

INTERVENTIONS:
Procedure: Stent placement — Surgeon may choose to use a single or double J ureteral stent (6- to 8.5-fr in size) or an alternative ureteral stent of the surgeon's choice.
  Arms: Stent vs No Stent
Drug: Alvimopan — Patient will receive alvimopan as a fixed 12-mg dose, with the first dose administered 0.5 to 5 h before the start of surgery; administration will be continued with twice daily oral doses postoperatively until hospital discharge or a maximum of 7 days (15 in-hospital doses).
  Arms: Alvimopan vs No Alvimopan

SUMMARY:
The purpose of this study is to look at two standard surgical techniques used during a radical cystectomy and see whether they influence outcomes such as length of stay in the hospital and infections after surgery. This trial will evaluate whether the following surgical methods influence outcomes:

A ureteral stent is a thin tube that is placed in the ureter to drain urine from the kidney. Ureteral stents are often used to promote urine drainage after radical cystectomy, but may come at risk of urinary tract infection.

Alvimopan is a standard drug used to promote return of bowel function following surgery. Doctors do not know whether alvimopan is beneficial in current clinical practice.

The surgeon will decide whether participants will receive a stent and/or alvimopan, but if they are unsure what the best approach is, a surgical technique has been assigned by chance to them.

ELIGIBILITY:
Inclusion Criteria:

Stent vs. no stent

* Patients aged ≥21 years who are scheduled to undergo radical cystectomy for treatment of bladder cancer with one of the consenting surgeons at MSK Alvimopan vs. no alvimopan
* Patients aged ≥21 years who are scheduled to undergo radical cystectomy for treatment of bladder cancer with one of the consenting surgeons at MSK

Exclusion Criteria:

Stent vs. no stent

* No exclusion criteria Alvimopan vs. no alvimopan
* Patients on chronic opioid therapy are ineligible to receive alvimopan and will be excluded from this cohort of the trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay (Alvimopan) | greater than 6 days
  it will define success for the intervention as a length of stay <6 days (6 days is the current median length of stay).
Symptomatic urinary tract infections (Stents) | within 30 days of surgery
  defined as the presence of signs or symptoms indicative of infection (fever, flank or abdominal pain, leukocytosis, radiographic imaging consistent with pyelonephritis) and a positive urine culture (>100,000 CFU pathogenic bacteria on an appropriately collected urine specimen).

CONTACTS AND LOCATIONS:
Overall Officials: Alvin Goh, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm